CLINICAL TRIAL: NCT00952380
Title: A THREE MONTH PROSPECTIVE OPEN LABEL STUDY OF THERAPY WITH FRAGMIN(REGISTERED) (DALTEPARIN SODIUM INJECTION) IN CHILDREN WITH VENOUS THROMBOEMBOLISM WITH OR WITHOUT MALIGNANCIES
Brief Title: Fragmin for the Treatment of Acute VTE in Pediatric Cancer Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FRAG-A001-201; A6301094 (Other: Alias Study Number); 2016-000394-21 (EudraCT Number)
Record Dates: First submitted 2009-08-04; First posted 2009-08-06 (Estimated); Results first posted 2019-04-16 (Actual); Last update posted 2019-04-16 (Actual); Status verified 2019-03

CONDITIONS: Venous Thromboembolism
Keywords: VTE
MeSH Terms: conditions — Venous Thromboembolism | interventions — Dalteparin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single Arm (Other): Single arm open-label
  Interventions: Drug: dalteparin

INTERVENTIONS:
Drug: dalteparin — dalteparin subcutaneous injection

SUMMARY:
Three month treatment of acute VTE with Fragmin in pediatric cancer patients

DETAILED DESCRIPTION:
Primary study objectives include are to determine the pharmacodynamic (PD) profiles for treatment doses of dalteparin in pediatric subjects of different ages with cancer and venous thromboembolism (VTE), using anti-Xa (Xa) levels and a population PD analysis methodology, and to determine the median dose required to achieve therapeutic anti- Xa levels (0.5 to 1.0 International Units [IU]/mL) based on subject age and weight.

ELIGIBILITY:
Inclusion Criteria:

-

Exclusion Criteria:

-

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 38 (Actual)
Dates: Start 2009-08 (Actual); Primary Completion 2018-03 (Actual); Study Completion 2018-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (26):
- United States (17):
  - Children's Hospital Colorado, Aurora, Colorado
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - Nemours Children's Clinic, Jacksonville, Florida
  - Wolfson Children's Hospital, Jacksonville, Florida
  - Investigational Drug Service Tampa General Hospital, Tampa, Florida
  - Tampa General Hospital Center of Research Excellence, Tampa, Florida
  - Tampa General Hospital, Tampa, Florida
  - University of South Florida, Tampa, Florida
  - St. Joseph's Children's Hospital of Tampa, Tampa, Florida
  - Children's Hospital of Michigan, Detroit, Michigan
  - Children's Mercy Hospitals and Clinics, Kansas City, Missouri
  - St. Jude Children's Research Hospital, Memphis, Tennessee
  - El Paso Children's Hospital, El Paso, Texas
  - Texas Tech University Health Sciences Center El Paso, El Paso, Texas
  - Texas Children's Cancer and Hematology Centers, Houston, Texas
  - Texas Children's Hospital Investigational Pharmacy Services, Houston, Texas
  - Texas Children's Hospital, Houston, Texas
- Norway (2):
  - Sykehusapoteket Oslo, Oslo
  - Oslo universitetssykehus HF, Oslo
- Russia (3):
  - FSBEI HE Kazan SMU of Minzdrav Russia, Kazan', Republic Tatarstan
  - SAHI "Children's Republican Clinical Hospital of the Ministry of, Kazan', Republic Tatarstan
  - SBHI of Moscow city Morozovskaya Children City Clinical Hospital of Moscow city, Moscow
- Slovenia (2):
  - Lekarna, Univerzitetni klinicni center Ljubljana, Ljubljana
  - Pediatricna klinika, Univerzitetni Klinicni Center Ljubljana, Ljubljana
- Spain (2):
  - Hospital HM Universitario Monteprincipe Servicio de Farmacia, Boadilla del Monte, Madrid
  - Hospital HM Universitario Monteprincipe, Boadilla del Monte, Madrid

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Hartman LR, Nurmeev I, Svirin P, Wolter KD, Yan JL, Jani D, Goldenberg NA, Sherman N. A phase 2 pharmacodynamic dose-finding, safety, and efficacy study of dalteparin for pediatric venous thromboembolism treatment in children with and without cancer. Pediatr Blood Cancer. 2022 Aug;69(8):e29764. doi: 10.1002/pbc.29764. Epub 2022 Jun 9. PMID 35678616
- [Derived] Damle B, Jen F, Sherman N, Jani D, Sweeney K. Population Pharmacokinetic Analysis of Dalteparin in Pediatric Patients With Venous Thromboembolism. J Clin Pharmacol. 2021 Feb;61(2):172-180. doi: 10.1002/jcph.1716. Epub 2020 Aug 21. PMID 32827160
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=FRAG-A001-201&StudyName=A%20Three%20Month%20Prospective%20Open%20Label%20Study%20Of%20Therapy%20With%20Fragmin%20%28registered%29%20%28dalteparin%20Sodium%20Injection%29%20In%20Children%20With%20Venous%20Thromboembolism%20With%20Or%20Without%20Malignancies
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=FRAG-A001-201&StudyName=A+Three+Month+Prospective+Open+Label+Study+Of+Therapy+With+Fragmin%28registered%29+%28dalteparin+Sodium+Injection%29+In+Children+With+Venous+Thromboembolism+With+Or+Without+Malignancies

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study was conducted in the 5 countries from 20 August 2009 to 20 March 2018. A total of 38 participants were enrolled. This study had dose adjustment (DA) phase (Day 1-7), pharmacodynamic (PD) phase (Day 8-14) and follow up (FU) phase (Day 15-104).
Groups:
- Dalteparin Sodium: Group 1 (>=0 to <8 Weeks): Participants aged greater than or equal to (>=) 0 to less than (<) 8 weeks were administered 125 international unit per kilogram (IU/kg) of dalteparin sodium injection subcutaneously twice daily from Day 1 to 7 in DA phase, Day 8 to 14 in PD phase and from Day 15 in FU phase (up to 104 days). Participants were to participate in the study for up to 104 days of study drug treatment to monitor the status of the qualifying venous thromboembolism (VTE). Participants were followed up for safety for up to 28 days after last dose of study drug (up to 132 days).
- Dalteparin Sodium: Group 2 (>=8 Weeks to <2 Years): Participants aged >=8 weeks to <2 years were administered 150 IU/kg of dalteparin sodium injection subcutaneously twice daily from Day 1 to 7 in DA phase, Day 8 to 14 in PD phase and from Day 15 in FU phase (up to 104 days). Participants were to participate in the study for up to 104 days of study drug treatment to monitor the status of the qualifying VTE. Participants were followed up for safety for up to 28 days after last dose of study drug (up to 132 days).
- Dalteparin Sodium: Group 3 (>=2 Years to <8 Years): Participants aged >=2 years to <8 years were administered 125 IU/kg of dalteparin sodium injection subcutaneously twice daily from Day 1 to 7 in DA phase, Day 8 to 14 in PD phase and from Day 15 in FU phase (up to 104 days). Participants were to participate in the study for up to 104 days of study drug treatment to monitor the status of the qualifying VTE. Participants were followed up for safety for up to 28 days after last dose of study drug (up to 132 days).
- Dalteparin Sodium: Group 4 (>=8 Years to <12 Years): Participants aged >=8 years to <12 years were administered 125 IU/kg of dalteparin sodium injection subcutaneously twice daily from Day 1 to 7 in DA phase, Day 8 to 14 in PD phase and from Day 15 in FU phase (up to 104 days). Participants were to participate in the study for up to 104 days of study drug treatment to monitor the status of the qualifying VTE. Participants were followed up for safety for up to 28 days after last dose of study drug (up to 132 days).
- Dalteparin Sodium: Group 5 (>=12 Years to <19 Years): Participants aged >=12 years to <19 years were administered 100 IU/kg of dalteparin sodium injection subcutaneously twice daily from Day 1 to 7 in DA phase, Day 8 to 14 in PD phase and from Day 15 in FU phase (up to 104 days). Participants were to participate in the study for up to 104 days of study drug treatment to monitor the status of the qualifying VTE. Participants were followed up for safety for up to 28 days after last dose of study drug (up to 132 days).
Period: Overall Study
Arm/Group | Dalteparin Sodium: Group 1 (>=0 to <8 Weeks) | Dalteparin Sodium: Group 2 (>=8 Weeks to <2 Years) | Dalteparin Sodium: Group 3 (>=2 Years to <8 Years) | Dalteparin Sodium: Group 4 (>=8 Years to <12 Years) | Dalteparin Sodium: Group 5 (>=12 Years to <19 Years)
Started | 1 | 2 | 8 | 7 | 20
Completed | 1 | 1 | 6 | 4 | 14
Not Completed | 0 | 1 | 2 | 3 | 6
Not completed — Other | 0 | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0 | 2
Not completed — Adverse Event | 0 | 1 | 0 | 0 | 3
Not completed — Physician Decision | 0 | 0 | 1 | 2 | 0
Not completed — Non-compliant to protocol | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: The safety analysis set included all the participants who received at least 1 dose of study drug.
Groups:
- Dalteparin Sodium: Group 1 (>=0 to <8 Weeks): Participants aged >= 0 to < 8 weeks were administered 125 IU/kg of dalteparin sodium injection subcutaneously twice daily from Day 1 to 7 in DA phase, Day 8 to 14 in PD phase and from Day 15 in FU phase (up to 104 days). Participants were to participate in the study for up to 104 days of study drug treatment to monitor the status of the qualifying VTE. Participants were followed up for safety for up to 28 days after last dose of study drug (up to 132 days).
- Total: Total of all reporting groups
Arm/Group | Dalteparin Sodium: Group 1 (>=0 to <8 Weeks) | Dalteparin Sodium: Group 2 (>=8 Weeks to <2 Years) | Dalteparin Sodium: Group 3 (>=2 Years to <8 Years) | Dalteparin Sodium: Group 4 (>=8 Years to <12 Years) | Dalteparin Sodium: Group 5 (>=12 Years to <19 Years) | Total
Number analyzed (Participants) | 1 | 2 | 8 | 7 | 20 | 38
Age, Continuous [Median (Full Range); unit: years] | 0.0684 [0.0684 to 0.0684] | 1.0569 [0.1999 to 1.9138] | 5.3676 [2.3409 to 7.3949] | 10.0287 [8.3833 to 11.8741] | 15.7208 [12.4682 to 18.7187] | 11.1577 [0.0684 to 18.7187]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 2 | 5 | 6 | 14
  Male | 1 | 1 | 6 | 2 | 14 | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 2 | 2 | 4 | 8
  Not Hispanic or Latino | 1 | 2 | 6 | 5 | 16 | 30
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 3 | 4 | 7
  White | 1 | 2 | 7 | 4 | 15 | 29
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 1 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Median Dose of Dalteparin Required to Achieve Prespecified Therapeutic Anti- Factor Xa Level
Description: Prespecified therapeutic anti-factor Xa level was 0.5-1.0 international unit per milliliter (IU/mL). Cumulative data of Day 1 to 7 has been reported.
Time Frame: 4 hours post-dose at each Day 1 to 7 in dose adjustment phase
Population: The pharmacodynamic (PD) analysis set included all participants who received at least 1 dose of study drug and achieved therapeutic range of anti-factor Xa during dose adjustment phase.
Measure: Median (Full Range); unit: IU/mL
Groups:
- Dalteparin Sodium: All Participants (>= 0 to < 19 Years): All participants who received dalteparin sodium injection, subcutaneously at a dose of 100 to 150 IU/kg twice daily from Day 1 to 7 in dose adjustment phase, Day 8-14 in PD phase and from Day 15 in follow up phase until bleeding necessitating or unexpected permanent discontinuation of anticoagulation therapy, unexpected thrombocytopenia and other adverse event necessitating discontinuation of study drug (up to a maximum of 104 days). Participants were followed up for safety for up to 28 days after last dose of study drug (up to 132 days).
Arm/Group | Dalteparin Sodium: All Participants (>= 0 to < 19 Years)
Number analyzed (Participants) | 34
IU/mL | 125 [99.1 to 213.5]

2. Secondary Outcome: Percentage of Participants Who Achieved Prespecified Therapeutic Anti- Factor Xa Levels
Description: Prespecified therapeutic anti-factor Xa level was 0.5-1.0 IU/mL. Percentage of participants who achieved the prespecified level during the dose adjustment phase were reported in this outcome measure.
Time Frame: Day 1 to 7 in dose adjustment phase
Population: Analysis population included all the participants who received at least 1 dose of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Dalteparin Sodium: Group 1 (>=0 to <8 Weeks) | Dalteparin Sodium: Group 2 (>=8 Weeks to <2 Years) | Dalteparin Sodium: Group 3 (>=2 Years to <8 Years) | Dalteparin Sodium: Group 4 (>=8 Years to <12 Years) | Dalteparin Sodium: Group 5 (>=12 Years to <19 Years)
Number analyzed (Participants) | 1 | 2 | 8 | 7 | 20
percentage of participants | 0 [0.00 to 97.50] | 100.0 [15.81 to 100.0] | 100.0 [63.06 to 100.0] | 100.0 [59.04 to 100.0] | 85.0 [62.11 to 96.79]

3. Secondary Outcome: Number of Participants With New or Progressive Symptomatic Venous Thromboembolism (VTE)
Description: Symptomatic VTE defined as new or progressive signs and symptoms as judged by the investigator including but not limited to: objective swelling, pain or tenderness, pitting edema, erythema or cyanosis. Progression of VTE: Progression of clot burden in terms of severity of occlusion, or involvement of new venous segments at any time after the initial diagnosis.
Time Frame: Baseline up to 28 days after the last dose of study drug (up to Day 132)
Population: The PD analysis set included all participants who received at least 1 dose of study drug and achieved therapeutic range of anti-factor Xa during dose adjustment phase. Data for this outcome measure (OM) was not planned to be collected and analyzed for age group of >=0 to <8 weeks.
Measure: Count of Participants; unit: Participants
Arm/Group | Dalteparin Sodium: Group 2 (>=8 Weeks to <2 Years) | Dalteparin Sodium: Group 3 (>=2 Years to <8 Years) | Dalteparin Sodium: Group 4 (>=8 Years to <12 Years) | Dalteparin Sodium: Group 5 (>=12 Years to <19 Years)
Number analyzed (Participants) | 2 | 8 | 7 | 17
Participants | 0 | 0 | 1 | 0

4. Secondary Outcome: Time to First Occurrence of Symptomatic Recurrent Venous Thromboembolism (VTE)
Description: It was defined as the time interval (in days) between date of first study treatment and date of documentation of first VTE. VTEs included both DVT and PE. DVT is a blood clot in the deep veins of the leg. If a DVT clot breaks off from a vein wall and flows towards the lungs and blocks some or all of the blood supply, it becomes PE. When a blood clot breaks, loose and travels in the blood, this is called VTE. VTE was confirmed by at least one radiographic test and was defined as any new or progressive VTE whose signs and symptoms (identified by the investigator) included: objective swelling or tenderness, pitting edema, erythema or cyanosis.
Time Frame: Baseline up to 28 days after the last dose of study drug (up to Day 132)
Population: The PD analysis set included all participants who received at least 1 dose of study drug and achieved therapeutic range of anti-factor Xa during dose adjustment phase.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Dalteparin Sodium: All Participants (>= 0 to < 19 Years)
Number analyzed (Participants) | 34
days | NA [NA to NA] — Median and 95% CI was not estimable due to the low number of participants who had VTE.

5. Secondary Outcome: Percentage of Participants With Clinical Response of Progression, Regression, Resolution and No Change in Venous Thromboembolism (VTE)
Description: VTEs included both DVT and PE. DVT is a blood clot in the deep veins of the leg. PE is a blood clot in the lungs. Clinical response of progression was defined as progression of clot burden in terms of severity of occlusion, or involvement of new venous segments at any time after the initial diagnosis. Clinical response of regression: Regressed clot burden utilizing the same imaging modality as the screening visit. Clinical response of resolution: Thrombus resolution of the qualifying event measured by repeat imaging at the end of study (EOS) visit.
Time Frame: Baseline up to 28 days after the last dose of study drug (up to Day 132)
Population: The PD analysis set included all participants who received at least 1 dose of study drug and achieved therapeutic range of anti-factor Xa during dose adjustment phase. Data for this OM was not planned to be collected and analyzed for age group of >=0 to <8 weeks.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Dalteparin Sodium: Group 2 (>=8 Weeks to <2 Years) | Dalteparin Sodium: Group 3 (>=2 Years to <8 Years) | Dalteparin Sodium: Group 4 (>=8 Years to <12 Years) | Dalteparin Sodium: Group 5 (>=12 Years to <19 Years)
Number analyzed (Participants) | 2 | 8 | 7 | 17
percentage of participants
  Progression | 0 [0.00 to 84.19] | 0 [0.00 to 36.94] | 0 [0.00 to 40.96] | 0 [0.00 to 19.51]
  Regression | 0 [0.00 to 84.19] | 12.5 [0.32 to 52.65] | 14.3 [0.36 to 57.87] | 29.4 [10.31 to 55.96]
  Resolution | 100.0 [15.81 to 100.0] | 62.5 [24.49 to 91.48] | 57.1 [18.41 to 90.10] | 58.8 [32.92 to 81.56]
  No Change | 0 [0.00 to 84.19] | 0 [0.00 to 36.94] | 14.3 [0.36 to 57.87] | 5.9 [0.15 to 28.69]

6. Secondary Outcome: Percentage of Participants With Major and Minor Bleeding Event
Description: A bleeding event was considered as major if it was clinically overt and satisfies 1 or more of the following criteria: fatal bleeding, bleeding accompanied by a decrease in hemoglobin of at least 2 grams per deciliter 24 hours, Overt bleeding deemed by the attending physician to necessitate permanent discontinuation of trial medication, Overt bleeding deemed by the attending physician to be unrelated to the participant's underlying condition and accompanied by blood product administration or bleeding occurred at a critical site (intraocular, intracranial, retroperitoneal). A bleeding event was considered as minor if it was clinically overt but not meeting the criteria for major or clinically relevant no major bleeding (bleeding resulting in any medical or surgical interventions but which did not meet the criteria for major bleeding).
Time Frame: Baseline up to 28 days after the last dose of study drug (up to Day 132)
Population: The safety analysis set included all the participants who received at least 1 dose of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Dalteparin Sodium: Group 1 (>=0 to <8 Weeks) | Dalteparin Sodium: Group 2 (>=8 Weeks to <2 Years) | Dalteparin Sodium: Group 3 (>=2 Years to <8 Years) | Dalteparin Sodium: Group 4 (>=8 Years to <12 Years) | Dalteparin Sodium: Group 5 (>=12 Years to <19 Years)
Number analyzed (Participants) | 1 | 2 | 8 | 7 | 20
percentage of participants
  Major Bleeding | 0 [0.00 to 97.50] | 50.0 [1.26 to 98.74] | 0 [0.00 to 36.94] | 0 [0.00 to 40.96] | 0 [0.00 to 16.84]
  Minor Bleeding | 0 [0.00 to 97.50] | 0 [0.00 to 84.19] | 50.0 [15.70 to 84.30] | 57.1 [18.41 to 90.10] | 40.0 [19.12 to 63.95]

7. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent were events between first dose of study drug and up to 28 days after the last dose of study drug (up to Day 132) that were absent before treatment or that worsened relative to pretreatment state. AEs included both SAEs and non-SAEs.
Time Frame: Baseline up to 28 days after the last dose of study drug (up to Day 132)
Population: The safety analysis set included all the participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Dalteparin Sodium: Group 1 (>=0 to <8 Weeks) | Dalteparin Sodium: Group 2 (>=8 Weeks to <2 Years) | Dalteparin Sodium: Group 3 (>=2 Years to <8 Years) | Dalteparin Sodium: Group 4 (>=8 Years to <12 Years) | Dalteparin Sodium: Group 5 (>=12 Years to <19 Years)
Number analyzed (Participants) | 1 | 2 | 8 | 7 | 20
Participants
  AEs | 1 | 2 | 7 | 7 | 19
  SAEs | 0 | 2 | 3 | 3 | 13

8. Secondary Outcome: Number of Participants With Laboratory Abnormalities
Description: Criteria:hematology:hemoglobin, hematocrit, erythrocytes less than(<)0.8*lower limit of normal(LLN), platelets <0.5*LLN >1.75*upper limit of normal (ULN),leukocytes <0.6* LLN >1.5* ULN, lymphocytes, lymphocytes/Leukocytes, neutrophils, neutrophils/leukocytes <0.8* LLN >1.2* ULN, basophils, basophils/leukocytes, eosinophils, eosinophils/leukocytes monocytes monocytes/leukocytes >1.2*ULN, activated partial thromboplastin time, prothrombin time, prothrombin international normalized ratio >1.1* ULN. Clinical chemistry: bilirubin >1.5*ULN, aspartate aminotransferase, alanine aminotransferase, lactate dehydrogenase, alkaline phosphatase >3.0*ULN, protein, albumin <0.8* LLN >1.2* ULN, blood urea nitrogen, creatinine >1.3* ULN, sodium <0.95*LLN >1.05*ULN, potassium, chloride, calcium, magnesium <0.9* LLN >1.1* ULN, phosphate <0.8* LLN >1.2* ULN, glucose <0.6*LLN >1.5*ULN, estimated(est) creatinine clearance, est GFR modified and bedside schwartz, >1.0* ULN. Urinalysis: creatinine >1.0*ULN.
Time Frame: Baseline up to 104 days
Population: The safety analysis set included all the participants who received at least 1 dose of study drug. Here, "Overall Number of Participants Analyzed" signifies participants who were evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Dalteparin Sodium: Group 1 (>=0 to <8 Weeks) | Dalteparin Sodium: Group 2 (>=8 Weeks to <2 Years) | Dalteparin Sodium: Group 3 (>=2 Years to <8 Years) | Dalteparin Sodium: Group 4 (>=8 Years to <12 Years) | Dalteparin Sodium: Group 5 (>=12 Years to <19 Years)
Number analyzed (Participants) | 1 | 2 | 8 | 7 | 19
Participants | 1 | 2 | 8 | 5 | 19

9. Secondary Outcome: Absolute Values of Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DSBP) in Participants
Time Frame: Baseline, Day 1, Day 2, Day 30, Day 60, Day 90
Population: The safety analysis set included all the participants who received at least 1 dose of study drug. Here "number analyzed" signifies the number of participants evaluable at specific time points.
Measure: Median (Full Range); unit: millimeters of mercury (mmHg)
Arm/Group | Dalteparin Sodium: Group 1 (>=0 to <8 Weeks) | Dalteparin Sodium: Group 2 (>=8 Weeks to <2 Years) | Dalteparin Sodium: Group 3 (>=2 Years to <8 Years) | Dalteparin Sodium: Group 4 (>=8 Years to <12 Years) | Dalteparin Sodium: Group 5 (>=12 Years to <19 Years)
Number analyzed (Participants) | 1 | 2 | 8 | 7 | 20
millimeters of mercury (mmHg)
  SBP: Baseline: number analyzed (Participants) | 1 | 1 | 6 | 3 | 12
  SBP: Baseline | 101.00 [101.00 to 101.00] | 50.00 [50.00 to 50.00] | 110.50 [95.00 to 119.00] | 96.00 [94.00 to 119.00] | 117.50 [97.00 to 140.00]
  SBP: Day 1: number analyzed (Participants) | 1 | 2 | 4 | 6 | 15
  SBP: Day 1 | 97.00 [97.00 to 97.00] | 105.50 [63.00 to 148.00] | 112.0 [100.00 to 137.00] | 111.00 [100.00 to 126.00] | 113.00 [92.00 to 130.00]
  SBP: Day 2: number analyzed (Participants) | 1 | 1 | 8 | 7 | 18
  SBP: Day 2 | 94.00 [94.00 to 94.00] | 75.00 [75.00 to 75.00] | 107.00 [90.0 to 128.0] | 112.00 [101.0 to 126.0] | 119.50 [98.0 to 158.0]
  SBP: Day 30: number analyzed (Participants) | 1 | 1 | 7 | 5 | 17
  SBP: Day 30 | 77.0 [77.00 to 77.00] | 77.00 [77.00 to 77.00] | 112.00 [100.00 to 123.00] | 109.00 [100.00 to 113.00] | 118.00 [95.00 to 133.00]
  SBP: Day 60: number analyzed (Participants) | 1 | 1 | 7 | 5 | 14
  SBP: Day 60 | 74.00 [74.0 to 74.0] | 102.00 [102.0 to 102.0] | 101.00 [91.0 to 124.0] | 118.00 [102.0 to 130.0] | 117.50 [102.0 to 134.0]
  SBP: Day 90: number analyzed (Participants) | 1 | 2 | 8 | 7 | 19
  SBP: Day 90 | 76.00 [76.0 to 76.0] | 105.00 [93.0 to 117.0] | 97.50 [90.0 to 105.0] | 116.00 [99.0 to 123.0] | 116.00 [89.0 to 151.0]
  DSBP: Baseline: number analyzed (Participants) | 1 | 1 | 6 | 3 | 12
  DSBP: Baseline | 60.00 [60.00 to 60.00] | 41.00 [41.00 to 41.00] | 66.00 [50.00 to 77.00] | 67.00 [60.00 to 75.00] | 65.00 [46.00 to 80.00]
  DSBP: Day 1: number analyzed (Participants) | 1 | 2 | 4 | 6 | 15
  DSBP: Day 1 | 61.00 [61.00 to 61.00] | 57.00 [41.00 to 73.00] | 65.50 [50.00 to 87.00] | 66.50 [54.00 to 81.00] | 64.00 [48.00 to 80.00]
  DSBP: Day 2: number analyzed (Participants) | 1 | 1 | 8 | 7 | 18
  DSBP: Day 2 | 48.00 [48.00 to 48.00] | 53.00 [53.00 to 53.00] | 60.50 [53.00 to 70.00] | 70.00 [65.00 to 79.00] | 65.00 [53.00 to 95.00]
  DSBP: Day 30: number analyzed (Participants) | 1 | 1 | 7 | 5 | 17
  DSBP: Day 30 | 53.00 [53.00 to 53.00] | 61.00 [61.00 to 61.00] | 64.00 [54.00 to 68.00] | 68.00 [53.00 to 71.00] | 69.00 [55.00 to 87.00]
  DSBP: Day 60: number analyzed (Participants) | 1 | 1 | 7 | 5 | 14
  DSBP: Day 60 | 51.00 [51.00 to 51.00] | 57.00 [57.00 to 57.00] | 60.00 [46.00 to 73.00] | 67.00 [59.00 to 70.00] | 67.00 [57.00 to 80.00]
  DSBP: Day 90: number analyzed (Participants) | 1 | 2 | 8 | 7 | 19
  DSBP: Day 90 | 53.00 [53.00 to 53.00] | 55.50 [51.00 to 60.00] | 60.50 [52.00 to 70.00] | 67.00 [56.00 to 80.00] | 69.00 [59.00 to 95.00]

10. Secondary Outcome: Absolute Values of Heart Rate (HR) and Pulse Rate (PR) of Participants
Description: Heart rate and pulse rate of participants were measured in terms of beats per minute.
Time Frame: Baseline, Day 1, Day 2, Day 30, Day 60, Day 90
Population: as for outcome 9
Measure: Median (Full Range); unit: beats per minute (bpm)
Arm/Group | Dalteparin Sodium: Group 1 (>=0 to <8 Weeks) | Dalteparin Sodium: Group 2 (>=8 Weeks to <2 Years) | Dalteparin Sodium: Group 3 (>=2 Years to <8 Years) | Dalteparin Sodium: Group 4 (>=8 Years to <12 Years) | Dalteparin Sodium: Group 5 (>=12 Years to <19 Years)
Number analyzed (Participants) | 1 | 2 | 8 | 7 | 20
beats per minute (bpm)
  HR: Baseline: number analyzed (Participants) | 1 | 1 | 4 | 0 | 5
  HR: Baseline | 148.00 [148.00 to 148.00] | 146.00 [146.00 to 146.00] | 115.00 [66.00 to 126.00] |  | 70.00 [52.00 to 84.00]
  HR: Day 1: number analyzed (Participants) | 1 | 1 | 1 | 0 | 7
  HR: Day 1 | 146.00 [146.00 to 146.00] | 142.00 [142.00 to 142.00] | 112.00 [112.00 to 112.00] |  | 85.00 [46.00 to 139.00]
  HR: Day 2: number analyzed (Participants) | 1 | 1 | 5 | 0 | 8
  HR: Day 2 | 136.00 [136.00 to 136.00] | 130.00 [130.00 to 130.00] | 114.00 [100.00 to 136.00] |  | 75.00 [56.00 to 124.00]
  HR: Day 30: number analyzed (Participants) | 1 | 1 | 4 | 0 | 8
  HR: Day 30 | 138.00 [138.00 to 138.00] | 130.00 [130.00 to 130.00] | 120.50 [100.00 to 124.00] |  | 87.50 [56.00 to 126.00]
  HR: Day 60: number analyzed (Participants) | 1 | 1 | 4 | 0 | 8
  HR: Day 60 | 132.00 [132.00 to 132.00] | 184.00 [184.00 to 184.00] | 120.00 [114.00 to 139.00] |  | 94.50 [56.00 to 134.00]
  HR: Day 90: number analyzed (Participants) | 1 | 1 | 4 | 0 | 8
  HR: Day 90 | 122.00 [122.00 to 122.00] | 134.00 [134.00 to 134.00] | 107.00 [96.00 to 116.00] |  | 80.00 [66.00 to 118.00]
  PR: Baseline: number analyzed (Participants) | 0 | 0 | 2 | 3 | 7
  PR: Baseline |  |  | 96.50 [68.00 to 125.00] | 114.00 [80.00 to 119.00] | 73.00 [67.00 to 150.00]
  PR: Day 1: number analyzed (Participants) | 0 | 1 | 3 | 6 | 8
  PR: Day 1 |  | 108.00 [108.00 to 108.00] | 121.00 [86.00 to 122.00] | 87.00 [76.00 to 120.00] | 94.50 [72.00 to 123.00]
  PR: Day 2: number analyzed (Participants) | 0 | 0 | 3 | 7 | 10
  PR: Day 2 |  |  | 117.00 [113.00 to 138.00] | 98.00 [84.00 to 127.00] | 93.00 [57.00 to 161.00]
  PR: Day 30: number analyzed (Participants) | 0 | 0 | 3 | 5 | 9
  PR: Day 30 |  |  | 88.00 [88.00 to 147.00] | 101.00 [90.00 to 150.00] | 102.00 [72.00 to 123.00]
  PR: Day 60: number analyzed (Participants) | 0 | 0 | 3 | 5 | 6
  PR: Day 60 |  |  | 88.00 [88.00 to 99.00] | 93.00 [75.00 to 108.00] | 95.00 [62.00 to 117.00]
  PR: Day 90: number analyzed (Participants) | 0 | 1 | 3 | 7 | 11
  PR: Day 90 |  | 140.00 [140.00 to 140.00] | 114.00 [113.00 to 120.00] | 96.00 [67.00 to 109.00] | 92.00 [74.00 to 124.00]

11. Secondary Outcome: Absolute Values of Height of Participants
Time Frame: Baseline, Day 1, Day 2, Day 30, Day 60, Day 90
Population: as for outcome 9
Measure: Median (Full Range); unit: centimeters (cm)
Arm/Group | Dalteparin Sodium: Group 1 (>=0 to <8 Weeks) | Dalteparin Sodium: Group 2 (>=8 Weeks to <2 Years) | Dalteparin Sodium: Group 3 (>=2 Years to <8 Years) | Dalteparin Sodium: Group 4 (>=8 Years to <12 Years) | Dalteparin Sodium: Group 5 (>=12 Years to <19 Years)
Number analyzed (Participants) | 1 | 2 | 8 | 7 | 20
centimeters (cm)
  Baseline: number analyzed (Participants) | 1 | 1 | 4 | 2 | 9
  Baseline | 54.00 [54.00 to 54.00] | 55.00 [55.00 to 55.00] | 110.00 [98.00 to 125.50] | 133.00 [126.00 to 140.00] | 166.00 [142.00 to 178.00]
  Day 1: number analyzed (Participants) | 1 | 0 | 3 | 2 | 11
  Day 1 | 54.00 [54.00 to 54.00] |  | 115.80 [98.00 to 118.00] | 134.00 [126.00 to 142.00] | 166.00 [113.50 to 184.00]
  Day 2: number analyzed (Participants) | 0 | 0 | 6 | 5 | 15
  Day 2 |  |  | 107.90 [89.50 to 120.00] | 142.00 [126.00 to 159.90] | 166.90 [113.60 to 189.00]
  Day 30: number analyzed (Participants) | 1 | 1 | 5 | 6 | 14
  Day 30 | 60.00 [60.00 to 60.00] | 56.60 [56.60 to 56.60] | 115.10 [89.50 to 124.50] | 140.30 [128.00 to 159.90] | 167.75 [113.90 to 184.00]
  Day 60: number analyzed (Participants) | 1 | 1 | 5 | 5 | 13
  Day 60 | 63.00 [63.00 to 63.00] | 60.00 [60.00 to 60.00] | 115.00 [90.00 to 124.50] | 139.70 [128.00 to 161.60] | 168.50 [114.20 to 183.60]
  Day 90: number analyzed (Participants) | 1 | 1 | 6 | 5 | 18
  Day 90 | 64.00 [64.00 to 64.00] | 61.00 [61.00 to 61.00] | 109.50 [91.50 to 127.00] | 140.70 [129.00 to 161.60] | 166.65 [115.00 to 184.00]

12. Secondary Outcome: Absolute Values of Weight of Participants
Time Frame: Baseline, Day 1, Day 2, Day 30, Day 60, Day 90
Population: as for outcome 9
Measure: Median (Full Range); unit: kilograms
Arm/Group | Dalteparin Sodium: Group 1 (>=0 to <8 Weeks) | Dalteparin Sodium: Group 2 (>=8 Weeks to <2 Years) | Dalteparin Sodium: Group 3 (>=2 Years to <8 Years) | Dalteparin Sodium: Group 4 (>=8 Years to <12 Years) | Dalteparin Sodium: Group 5 (>=12 Years to <19 Years)
Number analyzed (Participants) | 1 | 2 | 8 | 7 | 20
kilograms
  Baseline: number analyzed (Participants) | 1 | 1 | 6 | 3 | 9
  Baseline | 4.05 [4.05 to 4.05] | 3.93 [3.93 to 3.93] | 18.78 [12.80 to 34.70] | 36.60 [25.40 to 45.80] | 60.00 [48.00 to 86.90]
  Day 1: number analyzed (Participants) | 1 | 1 | 4 | 3 | 13
  Day 1 | 4.17 [4.17 to 4.17] | 4.04 [4.04 to 4.04] | 17.23 [13.40 to 21.20] | 37.00 [25.40 to 40.60] | 63.40 [19.60 to 95.20]
  Day 2: number analyzed (Participants) | 1 | 1 | 7 | 6 | 16
  Day 2 | 4.50 [4.50 to 4.50] | 4.15 [4.15 to 4.15] | 14.95 [11.90 to 34.70] | 39.35 [25.40 to 64.50] | 58.00 [19.70 to 89.80]
  Day 30: number analyzed (Participants) | 1 | 1 | 7 | 6 | 17
  Day 30 | 6.30 [6.30 to 6.30] | 4.56 [4.56 to 4.56] | 15.50 [13.00 to 37.20] | 39.20 [23.00 to 64.50] | 63.80 [21.80 to 91.70]
  Day 60: number analyzed (Participants) | 1 | 1 | 7 | 5 | 14
  Day 60 | 7.15 [7.15 to 7.15] | 4.60 [4.60 to 4.60] | 16.60 [12.70 to 37.20] | 38.30 [24.10 to 68.60] | 65.80 [22.70 to 90.80]
  Day 90: number analyzed (Participants) | 1 | 1 | 7 | 6 | 19
  Day 90 | 7.70 [7.70 to 7.70] | 4.70 [4.70 to 4.70] | 21.50 [14.00 to 38.50] | 39.30 [24.40 to 68.60] | 59.60 [22.60 to 89.80]

13. Secondary Outcome: Absolute Values of Respiratory Rate of Participants
Description: Respiratory rate was defined as the number of breaths per minute.
Time Frame: Baseline, Day 1, Day 2, Day 30, Day 60, Day 90
Population: as for outcome 9
Measure: Median (Full Range); unit: breaths per minute
Arm/Group | Dalteparin Sodium: Group 1 (>=0 to <8 Weeks) | Dalteparin Sodium: Group 2 (>=8 Weeks to <2 Years) | Dalteparin Sodium: Group 3 (>=2 Years to <8 Years) | Dalteparin Sodium: Group 4 (>=8 Years to <12 Years) | Dalteparin Sodium: Group 5 (>=12 Years to <19 Years)
Number analyzed (Participants) | 1 | 2 | 8 | 7 | 20
breaths per minute
  Baseline: number analyzed (Participants) | 1 | 1 | 6 | 3 | 12
  Baseline | 35.00 [35.00 to 35.00] | 25.00 [25.00 to 25.00] | 24.00 [18.00 to 24.00] | 20.00 [18.00 to 30.00] | 20.00 [17.00 to 36.00]
  Day 1: number analyzed (Participants) | 1 | 2 | 4 | 6 | 15
  Day 1 | 34.00 [34.00 to 34.00] | 36.00 [36.00 to 36.00] | 21.00 [20.00 to 24.00] | 18.00 [16.00 to 20.00] | 18.00 [16.00 to 30.00]
  Day 2: number analyzed (Participants) | 1 | 1 | 7 | 7 | 17
  Day 2 | 34.00 [34.00 to 34.00] | 34.00 [34.00 to 34.00] | 20.00 [18.00 to 24.00] | 20.00 [18.00 to 24.00] | 18.00 [16.00 to 24.00]
  Day 30: number analyzed (Participants) | 1 | 1 | 7 | 4 | 16
  Day 30 | 34.00 [34.00 to 34.00] | 36.00 [36.00 to 36.00] | 22.00 [16.00 to 28.00] | 22.00 [20.00 to 24.00] | 18.00 [16.00 to 32.00]
  Day 60: number analyzed (Participants) | 1 | 1 | 7 | 4 | 14
  Day 60 | 30.00 [30.00 to 30.00] | 36.00 [36.00 to 36.00] | 20.00 [16.00 to 24.00] | 20.00 [18.00 to 20.00] | 20.00 [16.00 to 30.00]
  Day 90: number analyzed (Participants) | 1 | 2 | 7 | 6 | 19
  Day 90 | 24.00 [24.00 to 24.00] | 34.00 [32.00 to 36.00] | 22.00 [20.00 to 24.00] | 20.00 [18.00 to 22.00] | 18.00 [12.00 to 28.00]

14. Secondary Outcome: Absolute Values of Body Temperature of Participants
Time Frame: Baseline, Day 1, Day 2, Day 30, Day 60, Day 90
Population: as for outcome 9
Measure: Median (Full Range); unit: degree celsius
Arm/Group | Dalteparin Sodium: Group 1 (>=0 to <8 Weeks) | Dalteparin Sodium: Group 2 (>=8 Weeks to <2 Years) | Dalteparin Sodium: Group 3 (>=2 Years to <8 Years) | Dalteparin Sodium: Group 4 (>=8 Years to <12 Years) | Dalteparin Sodium: Group 5 (>=12 Years to <19 Years)
Number analyzed (Participants) | 1 | 2 | 8 | 7 | 20
degree celsius
  Baseline: number analyzed (Participants) | 1 | 1 | 6 | 3 | 12
  Baseline | 36.60 [36.60 to 36.60] | 36.70 [36.70 to 36.70] | 36.50 [36.10 to 37.30] | 37.00 [36.20 to 37.20] | 36.80 [35.60 to 39.30]
  Day 1: number analyzed (Participants) | 1 | 2 | 4 | 6 | 15
  Day 1 | 36.70 [36.70 to 36.70] | 36.85 [36.70 to 37.00] | 36.80 [36.70 to 36.90] | 36.70 [36.00 to 37.00] | 36.80 [36.10 to 37.10]
  Day 2: number analyzed (Participants) | 1 | 1 | 8 | 7 | 18
  Day 2 | 36.90 [36.90 to 36.90] | 36.40 [36.40 to 36.40] | 36.70 [35.30 to 37.30] | 36.70 [36.60 to 36.80] | 36.70 [36.40 to 37.70]
  Day 30: number analyzed (Participants) | 1 | 1 | 7 | 5 | 17
  Day 30 | 36.50 [36.50 to 36.50] | 36.50 [36.50 to 36.50] | 36.60 [35.50 to 37.30] | 36.50 [36.40 to 38.60] | 36.70 [35.10 to 37.10]
  Day 60: number analyzed (Participants) | 1 | 1 | 7 | 5 | 13
  Day 60 | 36.60 [36.60 to 36.60] | 36.70 [36.70 to 36.70] | 36.80 [36.40 to 38.60] | 36.60 [35.60 to 36.90] | 36.60 [35.70 to 37.00]
  Day 90: number analyzed (Participants) | 1 | 2 | 8 | 7 | 19
  Day 90 | 36.70 [36.70 to 36.70] | 37.15 [36.70 to 37.60] | 36.75 [35.90 to 37.50] | 36.90 [36.70 to 38.40] | 36.80 [36.10 to 38.40]

15. Secondary Outcome: Absolute Values of Body Length of Participants
Time Frame: Baseline, Day 1, Day 2, Day 30, Day 60, Day 90
Population: as for outcome 9
Measure: Median (Full Range); unit: centimeter
Arm/Group | Dalteparin Sodium: Group 1 (>=0 to <8 Weeks) | Dalteparin Sodium: Group 2 (>=8 Weeks to <2 Years) | Dalteparin Sodium: Group 3 (>=2 Years to <8 Years) | Dalteparin Sodium: Group 4 (>=8 Years to <12 Years) | Dalteparin Sodium: Group 5 (>=12 Years to <19 Years)
Number analyzed (Participants) | 1 | 2 | 8 | 7 | 20
centimeter
  Baseline: number analyzed (Participants) | 1 | 1 | 1 | 0 | 1
  Baseline | 54 [54 to 54] | 55 [55 to 55] | 100 [100 to 100] |  | 172 [172 to 172]
  Day 1: number analyzed (Participants) | 1 | 1 | 0 | 0 | 1
  Day 1 | 54 [54 to 54] | 55 [55 to 55] |  |  | 135 [135 to 135]
  Day 2: number analyzed (Participants) | 1 | 1 | 2 | 0 | 1
  Day 2 | 56 [56 to 56] | 55.30 [55.30 to 55.30] | 104.75 [89.50 to 120] |  | 135 [135 to 135]
  Day 30: number analyzed (Participants) | 1 | 1 | 3 | 0 | 1
  Day 30 | 60 [60 to 60] | 56.60 [56.60 to 56.60] | 100 [89.50 to 124.5] |  | 135 [135 to 135]
  Day 60: number analyzed (Participants) | 1 | 1 | 3 | 0 | 1
  Day 60 | 63 [63 to 63] | 60 [60 to 60] | 103 [90 to 124.5] |  | 135 [135 to 135]
  Day 90: number analyzed (Participants) | 1 | 1 | 2 | 0 | 2
  Day 90 | 64 [64 to 64] | 61 [61 to 61] | 97.75 [91.50 to 104] |  | 151.75 [135 to 168.5]

16. Secondary Outcome: Number of Participants With Physical Examination Abnormalities of Participants
Description: Physical examinations included head, eyes, ears, nose, throat, neck, heart, chest, lungs, abdomen, extremities, skin, neurological status and general appearance. Abnormality in physical examination was based on investigator's discretion. Only those categories in which at least 1 participant had abnormality were reported.
Time Frame: Screening, Visit 2 (Baseline), Visit 3 (Day 1), Visit 4 (Day 2), Visit 5 (Day 30), Visit 6 (Day 60), Visit 7 (Day 90)
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | Dalteparin Sodium: Group 1 (>=0 to <8 Weeks) | Dalteparin Sodium: Group 2 (>=8 Weeks to <2 Years) | Dalteparin Sodium: Group 3 (>=2 Years to <8 Years) | Dalteparin Sodium: Group 4 (>=8 Years to <12 Years) | Dalteparin Sodium: Group 5 (>=12 Years to <19 Years)
Number analyzed (Participants) | 1 | 2 | 8 | 7 | 20
Participants
  Abdomen: Screening: number analyzed (Participants) | 1 | 2 | 7 | 7 | 19
  Abdomen: Screening | 0 | 1 | 2 | 0 | 2
  Abdomen: Visit 2: number analyzed (Participants) | 1 | 1 | 4 | 0 | 7
  Abdomen: Visit 2 | 0 | 0 | 2 |  | 0
  Abdomen: Visit 3: number analyzed (Participants) | 1 | 2 | 4 | 6 | 12
  Abdomen: Visit 3 | 0 | 1 | 1 | 0 | 2
  Abdomen: Visit 4: number analyzed (Participants) | 1 | 2 | 7 | 7 | 18
  Abdomen: Visit 4 | 0 | 0 | 1 | 1 | 3
  Abdomen: Visit 5: number analyzed (Participants) | 1 | 1 | 7 | 6 | 17
  Abdomen: Visit 5 | 0 | 0 | 0 | 1 | 4
  Abdomen: Visit 6: number analyzed (Participants) | 1 | 1 | 7 | 4 | 14
  Abdomen: Visit 6 | 0 | 0 | 0 | 1 | 1
  Abdomen: Visit 7: number analyzed (Participants) | 1 | 2 | 7 | 7 | 18
  Abdomen: Visit 7 | 0 | 1 | 0 | 1 | 3
  Chest: Screening: number analyzed (Participants) | 1 | 2 | 7 | 7 | 19
  Chest: Screening | 0 | 0 | 1 | 2 | 2
  Chest: Visit 2: number analyzed (Participants) | 1 | 1 | 4 | 0 | 7
  Chest: Visit 2 | 0 | 0 | 2 |  | 0
  Chest: Visit 3: number analyzed (Participants) | 1 | 2 | 4 | 5 | 12
  Chest: Visit 3 | 0 | 0 | 0 | 2 | 0
  Chest: Visit 4: number analyzed (Participants) | 1 | 2 | 7 | 6 | 18
  Chest: Visit 4 | 0 | 0 | 0 | 3 | 1
  Chest: Visit 5: number analyzed (Participants) | 1 | 1 | 7 | 5 | 17
  Chest: Visit 5 | 0 | 0 | 0 | 1 | 0
  Chest: Visit 6: number analyzed (Participants) | 1 | 1 | 7 | 3 | 14
  Chest: Visit 6 | 0 | 0 | 0 | 1 | 0
  Chest: Visit 7: number analyzed (Participants) | 1 | 2 | 7 | 6 | 18
  Chest: Visit 7 | 0 | 0 | 0 | 2 | 3
  Extremities: Screening: number analyzed (Participants) | 1 | 2 | 7 | 7 | 19
  Extremities: Screening | 0 | 0 | 0 | 4 | 10
  Extremities: Visit 2: number analyzed (Participants) | 1 | 1 | 4 | 0 | 7
  Extremities: Visit 2 | 0 | 0 | 1 |  | 1
  Extremities: Visit 3: number analyzed (Participants) | 1 | 2 | 4 | 6 | 12
  Extremities: Visit 3 | 0 | 0 | 1 | 3 | 3
  Extremities: Visit 4: number analyzed (Participants) | 1 | 2 | 7 | 7 | 17
  Extremities: Visit 4 | 0 | 0 | 0 | 4 | 8
  Extremities: Visit 5: number analyzed (Participants) | 1 | 1 | 7 | 6 | 16
  Extremities: Visit 5 | 0 | 0 | 0 | 1 | 3
  Extremities: Visit 6: number analyzed (Participants) | 1 | 1 | 7 | 4 | 14
  Extremities: Visit 6 | 0 | 0 | 0 | 1 | 2
  Extremities: Visit 7: number analyzed (Participants) | 1 | 2 | 7 | 7 | 18
  Extremities: Visit 7 | 0 | 0 | 0 | 2 | 2
  Eyes: Screening: number analyzed (Participants) | 1 | 1 | 5 | 0 | 8
  Eyes: Screening | 0 | 0 | 1 |  | 1
  Eyes: Visit 2: number analyzed (Participants) | 1 | 1 | 3 | 0 | 5
  Eyes: Visit 2 | 0 | 0 | 0 |  | 1
  Eyes: Visit 3: number analyzed (Participants) | 1 | 1 | 1 | 0 | 7
  Eyes: Visit 3 | 0 | 0 | 0 |  | 1
  Eyes: Visit 4: number analyzed (Participants) | 1 | 1 | 4 | 0 | 8
  Eyes: Visit 4 | 0 | 0 | 0 |  | 2
  Eyes: Visit 5: number analyzed (Participants) | 1 | 1 | 4 | 0 | 8
  Eyes: Visit 5 | 0 | 0 | 0 |  | 1
  Eyes: Visit 6: number analyzed (Participants) | 1 | 1 | 4 | 0 | 8
  Eyes: Visit 6 | 0 | 0 | 0 |  | 1
  Eyes: Visit 7: number analyzed (Participants) | 1 | 1 | 4 | 0 | 8
  Eyes: Visit 7 | 0 | 0 | 0 |  | 1
  Eyes, ears, nose, throat:Screening: number analyzed (Participants) | 0 | 1 | 2 | 7 | 11
  Eyes, ears, nose, throat:Screening | 0 | 1 | 1 | 0 | 2
  Eyes, ears, nose, throat: Visit 3: number analyzed (Participants) | 0 | 1 | 3 | 6 | 5
  Eyes, ears, nose, throat: Visit 3 |  | 0 | 1 | 0 | 1
  Eyes, ears, nose, throat: Visit 4: number analyzed (Participants) | 0 | 1 | 3 | 7 | 10
  Eyes, ears, nose, throat: Visit 4 |  | 0 | 0 | 0 | 2
  Eyes, ears, nose, throat: Visit 5: number analyzed (Participants) | 0 | 0 | 3 | 6 | 9
  Eyes, ears, nose, throat: Visit 5 |  |  | 0 | 0 | 3
  Eyes, ears, nose, throat: Visit 6: number analyzed (Participants) | 0 | 0 | 3 | 4 | 6
  Eyes, ears, nose, throat: Visit 6 |  |  | 2 | 0 | 1
  Eyes, ears, nose, throat: Visit 7: number analyzed (Participants) | 0 | 1 | 3 | 7 | 10
  Eyes, ears, nose, throat: Visit 7 |  | 0 | 1 | 0 | 2
  General appearance: Screening: number analyzed (Participants) | 1 | 2 | 7 | 7 | 19
  General appearance: Screening | 0 | 0 | 2 | 1 | 3
  General appearance: Visit 2: number analyzed (Participants) | 1 | 1 | 4 | 0 | 7
  General appearance: Visit 2 | 0 | 0 | 1 |  | 0
  General appearance: Visit 3: number analyzed (Participants) | 1 | 2 | 4 | 6 | 12
  General appearance: Visit 3 | 0 | 0 | 1 | 0 | 1
  General appearance: Visit 4: number analyzed (Participants) | 1 | 2 | 7 | 7 | 18
  General appearance: Visit 4 | 0 | 0 | 0 | 1 | 2
  General appearance: Visit 5: number analyzed (Participants) | 1 | 1 | 7 | 6 | 17
  General appearance: Visit 5 | 0 | 0 | 0 | 0 | 2
  General appearance: Visit 6: number analyzed (Participants) | 1 | 1 | 7 | 4 | 14
  General appearance: Visit 6 | 0 | 1 | 0 | 0 | 1
  General appearance: Visit 7: number analyzed (Participants) | 1 | 2 | 7 | 7 | 18
  General appearance: Visit 7 | 0 | 0 | 1 | 2 | 2
  Head: Screening: number analyzed (Participants) | 1 | 2 | 7 | 7 | 19
  Head: Screening | 0 | 0 | 1 | 1 | 4
  Head: Visit 3: number analyzed (Participants) | 1 | 2 | 4 | 6 | 12
  Head: Visit 3 | 0 | 0 | 1 | 0 | 2
  Head: Visit 4: number analyzed (Participants) | 1 | 2 | 7 | 7 | 18
  Head: Visit 4 | 0 | 0 | 1 | 0 | 5
  Head: Visit 5: number analyzed (Participants) | 1 | 1 | 7 | 6 | 17
  Head: Visit 5 | 0 | 0 | 1 | 1 | 4
  Head: Visit 6: number analyzed (Participants) | 1 | 1 | 7 | 4 | 14
  Head: Visit 6 | 0 | 0 | 1 | 1 | 3
  Head: Visit 7: number analyzed (Participants) | 1 | 2 | 7 | 7 | 18
  Head: Visit 7 | 0 | 0 | 1 | 1 | 5
  Heart: Screening: number analyzed (Participants) | 1 | 2 | 7 | 7 | 19
  Heart: Screening | 0 | 0 | 1 | 1 | 0
  Heart: Visit 3: number analyzed (Participants) | 1 | 2 | 4 | 6 | 12
  Heart: Visit 3 | 0 | 1 | 0 | 0 | 0
  Heart: Visit 4: number analyzed (Participants) | 1 | 2 | 7 | 7 | 18
  Heart: Visit 4 | 0 | 1 | 1 | 0 | 1
  Heart: Visit 7: number analyzed (Participants) | 1 | 2 | 7 | 7 | 18
  Heart: Visit 7 | 0 | 1 | 0 | 0 | 2
  Lungs: Screening: number analyzed (Participants) | 1 | 2 | 7 | 7 | 19
  Lungs: Screening | 0 | 0 | 0 | 1 | 0
  Lungs: Visit 4: number analyzed (Participants) | 1 | 2 | 7 | 7 | 18
  Lungs: Visit 4 | 0 | 0 | 0 | 0 | 1
  Lungs: Visit 6: number analyzed (Participants) | 1 | 1 | 7 | 4 | 14
  Lungs: Visit 6 | 0 | 0 | 0 | 0 | 1
  Lungs: Visit 7: number analyzed (Participants) | 1 | 2 | 7 | 7 | 18
  Lungs: Visit 7 | 0 | 0 | 0 | 0 | 1
  Neck: Screening: number analyzed (Participants) | 1 | 2 | 7 | 7 | 19
  Neck: Screening | 0 | 1 | 1 | 1 | 2
  Neck: Visit 4: number analyzed (Participants) | 1 | 2 | 7 | 5 | 18
  Neck: Visit 4 | 0 | 0 | 0 | 0 | 1
  Neurological: Screening: number analyzed (Participants) | 1 | 2 | 7 | 7 | 19
  Neurological: Screening | 0 | 0 | 2 | 0 | 0
  Neurological: Visit 2: number analyzed (Participants) | 1 | 1 | 4 | 0 | 7
  Neurological: Visit 2 | 0 | 0 | 1 |  | 0
  Neurological: Visit 3: number analyzed (Participants) | 1 | 2 | 4 | 6 | 12
  Neurological: Visit 3 | 0 | 0 | 1 | 0 | 0
  Neurological: Visit 4: number analyzed (Participants) | 1 | 2 | 7 | 6 | 18
  Neurological: Visit 4 | 0 | 0 | 0 | 0 | 1
  Neurological: Visit 5: number analyzed (Participants) | 1 | 1 | 7 | 6 | 17
  Neurological: Visit 5 | 0 | 0 | 0 | 0 | 1
  Neurological: Visit 7: number analyzed (Participants) | 1 | 2 | 7 | 7 | 18
  Neurological: Visit 7 | 0 | 1 | 0 | 0 | 0
  Nose: Screening: number analyzed (Participants) | 1 | 1 | 5 | 0 | 8
  Nose: Screening | 0 | 0 | 1 |  | 0
  Nose: Visit 2: number analyzed (Participants) | 1 | 1 | 3 | 0 | 5
  Nose: Visit 2 | 0 | 0 | 1 |  | 0
  Skin: Screening: number analyzed (Participants) | 1 | 2 | 7 | 7 | 19
  Skin: Screening | 1 | 1 | 1 | 3 | 5
  Skin: Visit 2: number analyzed (Participants) | 1 | 1 | 4 | 0 | 7
  Skin: Visit 2 | 1 | 0 | 0 |  | 1
  Skin: Visit 3: number analyzed (Participants) | 1 | 2 | 4 | 6 | 12
  Skin: Visit 3 | 1 | 1 | 1 | 1 | 3
  Skin: Visit 4: number analyzed (Participants) | 1 | 2 | 7 | 7 | 18
  Skin: Visit 4 | 0 | 1 | 2 | 2 | 6
  Skin: Visit 5: number analyzed (Participants) | 1 | 1 | 7 | 6 | 17
  Skin: Visit 5 | 0 | 0 | 2 | 2 | 7
  Skin: Visit 6: number analyzed (Participants) | 1 | 1 | 7 | 4 | 14
  Skin: Visit 6 | 0 | 0 | 0 | 2 | 5
  Skin: Visit 7: number analyzed (Participants) | 1 | 2 | 7 | 7 | 18
  Skin: Visit 7 | 0 | 1 | 1 | 3 | 4

17. Secondary Outcome: Time to First Occurrence of Major Bleeding Event
Description: Time to first occurrence of major bleeding event was defined as the time interval (in days) between date of first study treatment and date of documentation of first major bleeding event. A bleeding event was considered as major if it was clinically overt and satisfies 1 or more of the following criteria: fatal bleeding, bleeding accompanied by a decrease in hemoglobin of at least 2 grams per deciliter, overt bleeding deemed by the attending physician to necessitate permanent discontinuation of trial medication, overt bleeding deemed by the attending physician to be unrelated to the participant's underlying condition and accompanied by blood product administration, bleeding occurred at a critical site (intraocular, intracranial, retroperitoneal or intraspinal).
Time Frame: Baseline up to 28 days after the last dose of study drug (up to Day 132)
Population: The safety analysis set included all the participants who received at least 1 dose of study drug.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Dalteparin Sodium: All Participants (>= 0 to < 19 Years)
Number analyzed (Participants) | 38
days | NA [NA to NA] — Median and 95% CI was not estimable due to the low number of participants who had bleeding episodes.

18. Secondary Outcome: Percentage of Participants Who Remained Within Prespecified Therapeutic Anti-Factor Xa Levels at Day 30, 60 and 90 in Follow up Phase
Description: Prespecified therapeutic anti-factor Xa level was 0.5-1.0 IU/mL. The percentage of participants who had anti factor-Xa levels within the prespecified therapeutic range at Day 30, 60 and 90 during the follow up phase were reported in this outcome measure.
Time Frame: Day 30, Day 60, Day 90 in follow up phase
Population: PD analysis set included all participants who received at least 1 dose of study drug and achieved therapeutic range of anti-factor Xa during dose adjustment phase. Here, "number analyzed" signifies number of participants analyzed at specific time points. Data for this OM was not planned to be collected and analyzed for age group of >=0 to <8 weeks.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Dalteparin Sodium: Group 2 (>=8 Weeks to <2 Years) | Dalteparin Sodium: Group 3 (>=2 Years to <8 Years) | Dalteparin Sodium: Group 4 (>=8 Years to <12 Years) | Dalteparin Sodium: Group 5 (>=12 Years to <19 Years)
Number analyzed (Participants) | 2 | 8 | 7 | 17
percentage of participants
  Day 30: number analyzed (Participants) | 1 | 5 | 6 | 15
  Day 30 | 100.0 [2.50 to 100.0] | 100.0 [47.82 to 100.0] | 33.3 [4.33 to 77.72] | 93.3 [68.05 to 99.83]
  Day 60: number analyzed (Participants) | 1 | 5 | 4 | 11
  Day 60 | 100.0 [2.50 to 100.0] | 100.0 [47.82 to 100.0] | 75.0 [19.41 to 99.37] | 81.8 [48.22 to 97.72]
  Day 90: number analyzed (Participants) | 1 | 4 | 2 | 11
  Day 90 | 100.0 [2.50 to 100.0] | 100.0 [39.76 to 100.0] | 50.0 [1.26 to 98.74] | 72.7 [39.03 to 93.98]

19. Secondary Outcome: Percentage of Participants With Anti-Factor Xa Levels Outside the Prespecified Range at Day 30, 60 and 90 in Follow up Phase
Description: Prespecified therapeutic anti-factor Xa range was 0.5-1.0 IU/mL. The percentage of participants who had anti-factor Xa levels outside the prespecified therapeutic range at Day 30, 60 and 90 during the follow up phase were reported in this outcome measure.
Time Frame: Day 30, Day 60, Day 90 in follow-up phase
Population: as for outcome 18
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Dalteparin Sodium: Group 2 (>=8 Weeks to <2 Years) | Dalteparin Sodium: Group 3 (>=2 Years to <8 Years) | Dalteparin Sodium: Group 4 (>=8 Years to <12 Years) | Dalteparin Sodium: Group 5 (>=12 Years to <19 Years)
Number analyzed (Participants) | 2 | 8 | 7 | 17
percentage of participants
  Day 30: number analyzed (Participants) | 1 | 5 | 6 | 15
  Day 30 | 0 [0.00 to 97.50] | 0 [0.00 to 52.18] | 66.7 [22.28 to 95.67] | 6.7 [0.17 to 31.95]
  Day 60: number analyzed (Participants) | 1 | 5 | 4 | 11
  Day 60 | 0 [0.00 to 97.50] | 0 [0.00 to 52.18] | 25.0 [0.63 to 80.59] | 18.2 [2.28 to 51.78]
  Day 90: number analyzed (Participants) | 1 | 4 | 2 | 11
  Day 90 | 0 [0.00 to 97.50] | 0 [0.00 to 60.24] | 50.0 [1.26 to 98.74] | 27.3 [6.02 to 60.97]

20. Secondary Outcome: Maintenance Dose of Dalteparin Required to Achieve Prespecified Therapeutic Anti- Factor Xa Levels
Description: Prespecified therapeutic anti-factor Xa level was 0.5-1.0 IU/mL. Cumulative data for day 1 to 7 has been reported.
Time Frame: 4 hours post-dose at each Day 1 to 7 in dose adjustment phase
Population: PD analysis set. Here, "number analyzed" signifies the number of participants analyzed at specific time points. Data for this OM was not planned to be collected and analyzed for age group of >=0 to <8 weeks.
Measure: Mean (Standard Deviation); unit: IU/kg
Arm/Group | Dalteparin Sodium: Group 2 (>=8 Weeks to <2 Years) | Dalteparin Sodium: Group 3 (>=2 Years to <8 Years) | Dalteparin Sodium: Group 4 (>=8 Years to <12 Years) | Dalteparin Sodium: Group 5 (>=12 Years to <19 Years)
Number analyzed (Participants) | 2 | 8 | 7 | 17
IU/kg | 207.50 (8.485) | 141.85 (23.550) | 132.40 (12.934) | 115.06 (17.164)

21. Secondary Outcome: Time to Achieve Prespecified Therapeutic Anti- Factor Xa Levels
Description: Time to achieve the target range (prespecified therapeutic anti- factor Xa levels) was defined as the number of days from the first dose of study drug to the final dose that achieves the target anti-factor Xa level. Prespecified therapeutic anti-factor Xa level was 0.5-1.0 IU/mL. Cumulative data of Day 1 to 7 is reported.
Time Frame: Day 1 to 7 in dose adjustment phase
Population: PD analysis set included all participants who received at least 1 dose of study drug and achieved therapeutic range of anti-factor Xa during dose adjustment phase. Data for this OM was not planned to be collected and analyzed for age group of >=0 to <8 weeks.
Measure: Median (Full Range); unit: days
Arm/Group | Dalteparin Sodium: Group 2 (>=8 Weeks to <2 Years) | Dalteparin Sodium: Group 3 (>=2 Years to <8 Years) | Dalteparin Sodium: Group 4 (>=8 Years to <12 Years) | Dalteparin Sodium: Group 5 (>=12 Years to <19 Years)
Number analyzed (Participants) | 2 | 8 | 7 | 17
days | 4.5 [4 to 5] | 3.0 [1 to 7] | 2.0 [1 to 3] | 2.0 [1 to 4]

22. Secondary Outcome: Number of Dose Adjustments Required to Achieve Prespecified Therapeutic Anti-Xa Levels
Description: During dose adjustment phase, doses were adjusted according to prespecified therapeutic anti-Xa levels in order to achieve target prespecified therapeutic anti-factor Xa levels (0.5 to 1.0 IU/mL). Number of dose adjustments which were done within the specified time window of up to 4 hours post dose on all days (1 to 7) to achieve the prespecified therapeutic anti-Xa levels are reported.
Time Frame: 4 hours post-dose at each Day 1 to 7 in dose adjustment phase
Population: as for outcome 21
Measure: Median (Full Range); unit: dose adjustment
Arm/Group | Dalteparin Sodium: Group 2 (>=8 Weeks to <2 Years) | Dalteparin Sodium: Group 3 (>=2 Years to <8 Years) | Dalteparin Sodium: Group 4 (>=8 Years to <12 Years) | Dalteparin Sodium: Group 5 (>=12 Years to <19 Years)
Number analyzed (Participants) | 2 | 8 | 7 | 17
dose adjustment | 3.5 [3 to 4] | 0.5 [0 to 2] | 0.0 [0 to 1] | 0.0 [0 to 2]

23. Other Pre Specified Outcome: Total Body Clearance of Dalteparin
Description: Drug clearance is a quantitative measure of the rate at which a drug substance is removed from the blood (rate at which a drug is metabolized or eliminated by normal biological processes). Clearance obtained after intravenous infusion dose (apparent clearance) is influenced by the fraction of the dose absorbed.
Time Frame: 4 hours post-dose at each Day 1 to 7 in dose adjustment phase
Population: Data not reported for the endpoint, since the PK data was collected and analyzed in a pooled analysis, together with data from two external studies; the results of this pooled analysis will be reported separately.
Arm/Group | Dalteparin Sodium: All Participants (>= 0 to < 19 Years)
Number analyzed (Participants) | 0

24. Other Pre Specified Outcome: Volume of Distribution of Dalteparin
Description: Volume of distribution is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired blood concentration of a drug.
Time Frame: 4 hours post-dose at each Day 1 to 7 in dose adjustment phase
Population: as for outcome 23
Arm/Group | Dalteparin Sodium: All Participants (>= 0 to < 19 Years)
Number analyzed (Participants) | 0

25. Other Pre Specified Outcome: Absorption Rate Constant (Ka) of Dalteparin
Time Frame: 4 hours post-dose at each Day 1 to 7 in dose adjustment phase
Population: as for outcome 23
Arm/Group | Dalteparin Sodium: All Participants (>= 0 to < 19 Years)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Baseline up to 28 days after the last dose of study drug (up to Day 132)
Description: Same event may appear as both an adverse event (AE) and serious adverse event (SAE). However, what is presented are distinct events. An event may be categorized as serious in 1 participant and as non-serious in another, or a participant may have experienced both a serious and non-serious event.
Arm/Group | Dalteparin Sodium: Group 1 (>=0 to <8 Weeks) | Dalteparin Sodium: Group 2 (>=8 Weeks to <2 Years) | Dalteparin Sodium: Group 3 (>=2 Years to <8 Years) | Dalteparin Sodium: Group 4 (>=8 Years to <12 Years) | Dalteparin Sodium: Group 5 (>=12 Years to <19 Years)
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/2 | 0/8 | 0/7 | 1/20
Serious Adverse Events (participants affected / at risk) | 0/1 | 2/2 | 3/8 | 3/7 | 13/20
Other Adverse Events (participants affected / at risk) | 1/1 | 2/2 | 7/8 | 7/7 | 16/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dalteparin Sodium: Group 1 (>=0 to <8 Weeks) (N=1) | Dalteparin Sodium: Group 2 (>=8 Weeks to <2 Years) (N=2) | Dalteparin Sodium: Group 3 (>=2 Years to <8 Years) (N=8) | Dalteparin Sodium: Group 4 (>=8 Years to <12 Years) (N=7) | Dalteparin Sodium: Group 5 (>=12 Years to <19 Years) (N=20)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 1 | 3
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0
Pancytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 2
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Intestinal haematoma (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Mucosal inflammation (General disorders) | 0 | 0 | 0 | 0 | 2
Pain (General disorders) | 0 | 0 | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 0 | 1 | 1 | 3
Anaphylactic reaction (Immune system disorders) | 0 | 0 | 0 | 0 | 1
Drug hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 0 | 1
Bacterial infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Oral herpes (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 3
Respiratory syncytial virus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 2
Viral infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Vulvovaginal candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 5
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Malnutrition (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Seizure like phenomena (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 2
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 1
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 1
Thrombophlebitis superficial (Vascular disorders) | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dalteparin Sodium: Group 1 (>=0 to <8 Weeks) (N=1) | Dalteparin Sodium: Group 2 (>=8 Weeks to <2 Years) (N=2) | Dalteparin Sodium: Group 3 (>=2 Years to <8 Years) (N=8) | Dalteparin Sodium: Group 4 (>=8 Years to <12 Years) (N=7) | Dalteparin Sodium: Group 5 (>=12 Years to <19 Years) (N=20)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 3 | 1 | 2
Coagulopathy (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 3
Pancytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 2 | 0 | 1
Tachycardia (Cardiac disorders) | 0 | 1 | 2 | 2 | 0
Cerumen impaction (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1
Dry eye (Eye disorders) | 0 | 0 | 0 | 1 | 1
Eye swelling (Eye disorders) | 0 | 0 | 0 | 0 | 1
Ocular hyperaemia (Eye disorders) | 0 | 0 | 0 | 1 | 0
Photophobia (Eye disorders) | 0 | 0 | 1 | 0 | 0
Vision blurred (Eye disorders) | 0 | 0 | 0 | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Abdominal tenderness (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Anal fissure (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Chapped lips (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Cheilitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 3 | 1 | 1
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Erosive oesophagitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 1 | 0
Haematoma (Vascular disorders) | 0 | 0 | 1 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 1 | 0 | 2
Vein disorder (Vascular disorders) | 0 | 0 | 1 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0
Drug hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 0 | 1
Hypocomplementaemia (Immune system disorders) | 0 | 0 | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1
Mental disorder (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
Leukocyturia (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
Vulvovaginal pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1
Gastrointestinal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Gingival bleeding (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1
Haematemesis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1
Intestinal dilatation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Intra-abdominal haematoma (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Lip dry (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Lip haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Mouth ulceration (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 2 | 1 | 0
Oesophageal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Perianal erythema (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Proctalgia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 2
Vomiting (Gastrointestinal disorders) | 0 | 2 | 1 | 2 | 1
Asthenia (General disorders) | 0 | 1 | 0 | 0 | 0
Catheter site bruise (General disorders) | 0 | 0 | 0 | 0 | 1
Catheter site haematoma (General disorders) | 0 | 0 | 0 | 0 | 1
Catheter site pain (General disorders) | 0 | 0 | 0 | 1 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 2
Gait disturbance (General disorders) | 0 | 0 | 1 | 0 | 0
Infusion site bruising (General disorders) | 0 | 0 | 0 | 0 | 1
Infusion site haemorrhage (General disorders) | 0 | 0 | 0 | 0 | 1
Injection site bruising (General disorders) | 0 | 1 | 2 | 4 | 8
Injection site haematoma (General disorders) | 0 | 0 | 1 | 0 | 1
Injection site haemorrhage (General disorders) | 0 | 0 | 0 | 1 | 1
Injection site mass (General disorders) | 0 | 0 | 1 | 0 | 0
Injection site nodule (General disorders) | 0 | 0 | 0 | 1 | 1
Injection site pain (General disorders) | 0 | 0 | 0 | 0 | 4
Localised oedema (General disorders) | 0 | 0 | 0 | 0 | 1
Mucosal haemorrhage (General disorders) | 0 | 0 | 1 | 0 | 0
Mucosal inflammation (General disorders) | 0 | 0 | 1 | 1 | 2
Nodule (General disorders) | 0 | 0 | 0 | 1 | 0
Oedema peripheral (General disorders) | 0 | 0 | 0 | 2 | 1
Pain (General disorders) | 0 | 0 | 0 | 2 | 1
Pyrexia (General disorders) | 0 | 1 | 2 | 2 | 2
Swelling (General disorders) | 0 | 0 | 0 | 0 | 1
Bone contusion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 2 | 3
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Refractoriness to platelet transfusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Catheter site inflammation (General disorders) | 0 | 0 | 0 | 1 | 0
Aspergillus infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Bacterial infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Bacteriuria (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Clostridium difficile colitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Clostridium difficile infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Conjunctivitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Genitourinary tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Influenza (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Infusion site cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Paronychia (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Rhinitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Rhinovirus infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Sinusitis bacteria (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Skin infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Stoma site cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Vaginal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Viral diarrhoea (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Viral infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Fluid overload (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Acanthosis nigricans (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 2
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 1
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 1
Pain of skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 1
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Red man syndrome (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Skin discolouration (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Skin disorder (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Skin induration (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Urticaria contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 3
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 4
Pharyngeal erythema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0 | 0
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Altered state of consciousness (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Ataxia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 2
Headache (Nervous system disorders) | 0 | 0 | 2 | 2 | 2
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Neuralgia (Nervous system disorders) | 0 | 0 | 1 | 0 | 1
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 0 | 1 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Activated partial thromboplastin time prolonged (Investigations) | 0 | 1 | 2 | 0 | 2
Alanine aminotransferase increased (Investigations) | 1 | 0 | 0 | 1 | 2
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 1 | 2
Aspergillus test positive (Investigations) | 0 | 0 | 0 | 0 | 1
Blood calcium increased (Investigations) | 0 | 1 | 0 | 0 | 0
Blood fibrinogen decreased (Investigations) | 0 | 0 | 0 | 0 | 1
Blood fibrinogen increased (Investigations) | 0 | 0 | 0 | 0 | 1
Blood lactate dehydrogenase increased (Investigations) | 0 | 0 | 1 | 0 | 0
Blood urea increased (Investigations) | 0 | 1 | 0 | 0 | 0
Body temperature increased (Investigations) | 0 | 1 | 0 | 0 | 0
C-reactive protein increased (Investigations) | 0 | 0 | 0 | 0 | 1
Haematocrit decreased (Investigations) | 0 | 0 | 0 | 0 | 1
Haemoglobin decreased (Investigations) | 0 | 0 | 0 | 2 | 1
Hepatitis A virus test positive (Investigations) | 0 | 0 | 0 | 0 | 1
International normalised ratio increased (Investigations) | 0 | 0 | 0 | 0 | 1
Lymphocyte count decreased (Investigations) | 0 | 0 | 0 | 0 | 1
Neutrophil count decreased (Investigations) | 0 | 0 | 0 | 1 | 1
Platelet count decreased (Investigations) | 0 | 0 | 0 | 2 | 1
Platelet count increased (Investigations) | 1 | 0 | 0 | 0 | 0
Prothrombin time prolonged (Investigations) | 0 | 0 | 0 | 0 | 2
Transaminases increased (Investigations) | 0 | 0 | 0 | 2 | 0
Weight decreased (Investigations) | 0 | 1 | 0 | 0 | 1
White blood cell count decreased (Investigations) | 0 | 0 | 0 | 1 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 2
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 1
Magnesium deficiency (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 2
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2016-10-18): https://cdn.clinicaltrials.gov/large-docs/80/NCT00952380/Prot_000.pdf
  • Statistical Analysis Plan (2015-11-18): https://cdn.clinicaltrials.gov/large-docs/80/NCT00952380/SAP_001.pdf